CLINICAL TRIAL: NCT03857243
Title: Dual Transcranial Direct Current Stimulation (dTDCS)-Enhanced Therapy After Hemorrhagic Strokes and VEGF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to administrative difficulties caused by PI change.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14GRNT18690039; STU 012014-028 (Other: IRB University of Texas Southwestern Medical Center)
Record Dates: First submitted 2017-06-21; First posted 2019-02-27 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Hemorrhagic Stroke; Hemiparesis
MeSH Terms: conditions — Hemorrhagic Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dTDCS plus physical therapy (Experimental): active dual transcranial direct current stimulation (TDCS) arm (M1-M1)
  Interventions: Device: dual transcranial direct current stimulation
- Sham dTDCS plus physical therapy (Placebo Comparator): Non-effective dose dual TDCS stimulation arm, identical with intervention arm except for the stimulation intensity/duration used.
  Interventions: Device: dual transcranial direct current stimulation

INTERVENTIONS:
Device: dual transcranial direct current stimulation — Mild, non-invasive battery powered direct current applied to the head over the motor areas. No shaving or invasive procedures needed.
  Other Names: dtDCS,; dual tDCS

SUMMARY:
This study will evaluate the feasibility of dual tDCS to improve arm motor function in chronic stroke patients. In addition it will collect pilot data on the blood biomarkers associated with treatment effect.

DETAILED DESCRIPTION:
The proposed, increased intensity dtDCS is a new, economical, noninvasive stimulation approach that has the potential for large-scale clinical application. Dual tDCS, in conjunction with physical and occupational therapy, is not only more effective in enhancing motor performance and cortical plasticity compared to sham, but approximately 50% more effective than cathodal or anodal stimulation in healthy subjects and after stroke. However, it will only be clinically useful and important if the beneficial effects persist over time in a wider stroke patient population. Improvement in inter-hemispheric balance, through an activation shift toward the affected hemisphere and clinical improvement in response to tDCS has been reported previously in small studies. Hemorrhagic stroke patients have not been evaluated.

The investigators will study rehabilitation associated cortical plasticity at a cellular level to gain insight into the neural substrates underlying the clinical improvement. There are no prior studies investigating the potential of VEGF polymorphisms to contribute to rehabilitative treatment-induced functional recovery in humans. The investigators expect that patients with VEGF genotype 2578A/A will recover less then subjects without this polymorphism. Since in animal models VEGF and BDNF have a complimentary role, VEGF polymorphism may explain some of the variability in strength of association between BDNF polymorphism Val66Met and recovery. This novel pilot study measures both the genetic and physiologic expression of multiple growth factors - before and after a promising new therapy regimen - to better understand the contribution of growth factors to long-term plasticity and functional recovery. If VEGF serum levels elevate with clinical improvement, then this may identify a new indicator of treatment efficacy that can be collected noninvasively and with little cost. The results will provide guidance for new inclusion/exclusion criteria for clinical studies based on genetic markers, as well as uncover the potential for new therapeutic strategies to enhance treatment efficacy by augmenting VEGF during rehabilitation with FDA-approved strategies currently in clinical trials for other conditions (NIH Clinical Trials Registry: NCT01384162, NCT00620217, and NCT00744315).

ELIGIBILITY:
Inclusion Criteria:

1. Patients (18-85 yo) with arm weakness (uFM <60) as a result of an ICH and no history of other neurologic or psychiatric illness that are able to activate wrist flexors (> MRC 1);
2. Patients with symptomatic ICH >5 months before enrollment;
3. Ashworth spasticity score <3.

Exclusion Criteria:

1. Patients with severe uncontrolled medical problems,
2. Patients with subarachnoid, subdural or epidural hemorrhage;
3. Patients with unstable cardiac arrhythmia;
4. Patients with contraindication to tDCS stimulation;
5. Patients who are not available for follow-up or unable to follow study procedures;
6. Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects were found not eligible for participation after signing consent.
Period: Overall Study
Arm/Group | dTDCS Plus Physical Therapy | Sham dTDCS Plus Physical Therapy
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dTDCS Plus Physical Therapy | Sham dTDCS Plus Physical Therapy | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Nonhispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: any adverse events that might be related to study procedures
Time Frame: enrollment to 3 month followup
Measure: Number; unit: number of events
Arm/Group | dTDCS Plus Physical Therapy | Sham dTDCS Plus Physical Therapy
Number analyzed (Participants) | 1 | 1
number of events | 0 | 0

2. Primary Outcome: Upper Extremity Fugl-Meyer Score
Description: Upper extremity motor impairment scale. Scale ranges from 0 (worst, can not perform any tasks) to 66 ( performs all tasks fully).
Time Frame: change between before and 3 months follow-up
Population: One subject finished the treatment, statistical analysis was not performed
Arm/Group | dTDCS Plus Physical Therapy | Sham dTDCS Plus Physical Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Wolf Motor Function Test
Description: Timed performance of 15 functional upper extremity tasks, 0-120 seconds, and 2 strength measures.
  WMFT time measurements are calculated as the arithmetic mean of rate of performance, where we calculate "how many times would a person have completed the task, had he or she been performing it continuously for 60 seconds". Therefore the results have a minimum score of 0, where the subject could not perform any of the tasks, and no pre-defined maximum score, the higher the rate score the faster the subject was able to perform the tasks. ( see Hodics et al.,2013)
Time Frame: change between before and at 3 months follow-up
Population: One subject finished the treatment, statistical analysis was not performed
Arm/Group | dTDCS Plus Physical Therapy | Sham dTDCS Plus Physical Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | dTDCS Plus Physical Therapy | Sham dTDCS Plus Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Early termination due to PI relocation, low recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No